CLINICAL TRIAL: NCT01856257
Title: Steroid and Tacrolimus Avoidance Using NULOJIX® (Belatacept) in Renal Transplantation (CTOT-16)
Brief Title: Open-Label Phase 2 Trial of a Steroid-Free, CNI-Free, Belatacept-Based Immunosuppressive Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety: Stopping rule not met.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-16
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Primary Renal Allograft Candidate; Kidney Transplantation
Keywords: Kidney Transplantation; Transplantation; NULOJIX; belatacept; chronic immunosuppression
MeSH Terms: interventions — Antilymphocyte Serum; thymoglobulin; Abatacept; Methylprednisolone; Basiliximab; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thymoglobulin®+tacrolimus+MMF (Active Comparator): Induction with Thymoglobulin®, methylprednisolone, and maintenance immunosuppression with tacrolimus and mycophenolate mofetil (MMF)
  Interventions: Biological: Anti-thymocyte Globulin (Rabbit); Drug: methylprednisolone; Drug: mycophenolate mofetil; Drug: tacrolimus
- Thymoglobulin®+belatacept+MMF (Experimental): Induction with Thymoglobulin®, methylprednisolone, and maintenance with belatacept and mycophenolate mofetil (MMF)
  Interventions: Biological: Anti-thymocyte Globulin (Rabbit); Biological: belatacept; Drug: methylprednisolone; Drug: mycophenolate mofetil
- Basiliximab+20 weeks of tacrolimus+MMF + belatacept (Experimental): Induction basiliximab and methylprednisolone, administration of NULOJIX® (belatacept) 24 hours post reperfusion (+/-12 hrs); maintenance immunosuppression with 1. )20 week course of Prograf® (tacrolimus) or equivalent 2.) CellCept® (mycophenolate mofetil- MMF), or Myfortic® (mycophenolate sodium), or equivalent.
  Subjects participating in this arm may have tacrolimus reinstated, at a dose to be determined by the site investigator, if any of the following events occur: 1 - An acute rejection episode 2- Request of the subject or site Investigator.
  Interventions: Biological: belatacept; Drug: methylprednisolone; Biological: basiliximab; Drug: mycophenolate mofetil; Drug: tacrolimus

INTERVENTIONS:
Biological: Anti-thymocyte Globulin (Rabbit) — The target dosage is 6mg/kg total over 3 to 4 days. The recommended route of administration is intravenous infusion using a high-flow vein.
  Other Names: Thymoglobulin®; ATG (Rabbit)
  Arms: Thymoglobulin®+belatacept+MMF; Thymoglobulin®+tacrolimus+MMF
Biological: belatacept — Participants will receive belatacept at a dose of 10mg/kg up on day 1, 5, 14, 28, 56 and 84. After 84 days, subjects will receive a maintenance dose of 5 mg/kg every 4 weeks until completion of the trial.
  Other Names: NULOJIX®
  Arms: Basiliximab+20 weeks of tacrolimus+MMF + belatacept; Thymoglobulin®+belatacept+MMF
Drug: methylprednisolone — Methylprednisolone will be administered at a target dose of 500 mg beginning on the day of transplant, and tapered to 250 mg day 1 post-transplant, 125 mg day 2 post-transplant, 60 mg day 3 post-transplant, 30 mg day 4 post-transplant and day 5 post-transplant 0 mg if therapeutic tacrolimus level achieved for groups 1 and 3.
  Other Names: Medrol®
Biological: basiliximab — Basiliximab will be administered in two doses of 20 mg each.
  Other Names: Simulect®
  Arms: Basiliximab+20 weeks of tacrolimus+MMF + belatacept
Drug: mycophenolate mofetil — Mycophenolate Mofetil will be administered at a target dose of 1000 mg orally twice a day. Myfortic® (mycophenolate sodium) may be used as a replacement for MMF. Mycophenolate sodium will be dosed at 720 mg PO BID. Mycophenolate sodium will be adjusted based on clinical complications.
  Other Names: MMF; CellCept®; mycophenolate acid
Drug: tacrolimus — The site investigator will identify a starting tacrolimus dose at their discretion, in order to achieve the target trough levels, no later than 5 days post-transplantation. The dose will be adjusted to 5-8ng/ml for the active comparator arm (thymoglobulin + tacrolimus + MMF arm) or tapered off in the experimental arm (basiliximab + 20 weeks of tacrolimus + MMF + belatacept).
  Other Names: Prograf®
  Arms: Basiliximab+20 weeks of tacrolimus+MMF + belatacept; Thymoglobulin®+tacrolimus+MMF

SUMMARY:
The primary objective is to evaluate a NULOJIX® (belatacept) based regimens as a means of improving long-term graft function without increasing the risks of immunologic graft injury by avoiding both calcineurin inhibitors (CNIs) and corticosteroids.

DETAILED DESCRIPTION:
Taking standard anti-rejection medications for a long time can cause serious side effects, including kidney damage. Transplant recipients have to take anti-rejection medications to prevent their immune system (the body's natural defense system against illness) from rejecting their new kidney. Most patients who receive a kidney transplant must take these anti-rejection medications for the rest of their lives, or for as long as the kidney continues to work.

The purpose of this study is to determine if NULOJIX® (belatacept), will minimize serious long term side effects seen with anti-rejection medications while still protecting the transplanted kidney from damage. The researchers also want to learn more about the safety of this treatment and the long term health of the transplanted kidney.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18-65 years of age at the time of enrollment;
* Ability to understand and provide written informed consent;
* Candidate for primary renal allograft from either living or deceased donor;
* No known contraindications to study therapy using NULOJIX® (belatacept);
* Female participants of childbearing potential must have a negative pregnancy test upon study entry;
* Participants with reproductive potential must agree to use an appropriate method(s) of birth control as outlined in the CellCept® , Myfortic® or generic package labeling during participation in the study and for 4 months following completion of the study;
* No donor specific antibodies prior to transplant that are considered to be of clinical significance by the site investigator;
* Negative crossmatch or Panel Reactive Antibodies (PRA) of 0% on historic and current sera, as determined by each participating study center;
* A documented negative tuberculosis (TB) test within the 6 months prior to transplant. If documentation is not present at the time of transplantation, and the subject does not have any risk factors for TB, a TB-specific interferon gamma release assay (IGRA) may be performed.

Exclusion Criteria:

* Need for multi-organ transplant;
* Recipient of previous organ transplant;
* Epstein-Barr Virus (EBV) seronegative (or unknown) recipients;
* Active infection including hepatitis B, hepatitis C, or human Immunodeficiency Virus (HIV);
* Individuals who have required treatment with prednisone or other immunosuppressive drugs within 1 year prior to transplant;
* Individuals undergoing transplant using organs from extended criteria donor (ECD) or donation after cardiac death (DCD) donors;
* Histocompatibility antigen (HLA) identical living donors;
* Individuals at significant risk of early recurrence of the primary renal disease including focal segmental glomerulosclerosis (FSGS) and membranoproliferative glomerulonephritis (MPGN) type 2 or any other disease that in the opinion of the investigator is at increased likelihood of recurrence and which may result in rapid decline in renal function;
* Known history of thrombotic events or risk factors, including any of the following:

  * Factor V Leiden, elevated homocysteine, positive lupus anticoagulant, elevated anticardiolipin antibody, heparin-induced thrombocytopenia,
  * A family history of a heritable thrombotic condition,
  * Recurrent deep vein thrombosis (DVT) or pulmonary emboli (PE),
  * Unexplained stillborn infant or recurrent spontaneous abortion or other congenital or acquired thrombotic disorder.

At the discretion of the investigator, a history of thrombosis of a dialysis access graft, fistula, or indwelling catheter/device may not be considered an exclusion criterion.

* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements;
* Use of investigational drugs within 4 weeks of enrollment;
* Known hypersensitivity to mycophenolate mofetil (MMF)or any of the drug's components;
* Administration of live attenuated vaccine(s) within 8 weeks of enrollment;
* Blood type A2 and A2B donors into blood type B recipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Newell, MD, PhD, Principal Investigator — Emory University; Roslyn B. Mannon, M.D., Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Participant level data access and additional relevant materials will be made available upon completion of the trial.
Supporting Information: Study Protocol
Time Frame: After completion of the trial, within 24 months status post database lock.
Access Criteria: Study Accession ID: SDY1434
  Registration is available for the Immunology Database and Analysis Portal (ImmPort) at: https://www.immport.org/registration and submit a rationale for the purpose of requesting study data access.
  ImmPort is a long-term archive of clinical and mechanistic data, a National Institute of Allergy and Infectious Diseases Division of Allergy, Immunology and Transplantation (NIAID DAIT)-funded data repository. This archive is in support of the NIH mission to share data with the public. Data shared through ImmPort is provided by NIH-funded programs, other research organizations and individual scientists, ensuring these discoveries will be the foundation of future research.
URL: https://www.immport.org/shared/study/SDY1434

REFERENCES:
- [Result] Mannon RB, Armstrong B, Stock PG, Mehta AK, Farris AB, Watson N, Morrison Y, Sarwal M, Sigdel T, Bridges N, Robien M, Newell KA, Larsen CP. Avoidance of CNI and steroids using belatacept-Results of the Clinical Trials in Organ Transplantation 16 trial. Am J Transplant. 2020 Dec;20(12):3599-3608. doi: 10.1111/ajt.16152. Epub 2020 Jul 13. PMID 32558199
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three sites in the United States recruited and enrolled 71 participants into this trial.
Groups:
- Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac: Induction:
  Methylprednisolone (MEDROL) was administered at a dose of 500mg on the day of transplant, and tapered to 250 mg on day 1, 125 mg on day 2, 60 mg on day 3, 30 mg on day 4, and 0 mg on day 5.
  Thymoglobulin via intravenous infusion was administered at a target dose of 6 mg/kg over 3 to 4 days.
  Maintenance:
  Mycophenolate Mofetil (MMF) or equivalent was administered at a target dose of 1000 mg PO or IV BID starting on the day of transplant or day 1.
  The site investigator determined the starting dose. The first tacrolimus (tac) dosing was administered on the day of transplant or day 1 and was adjusted to achieve a target trough of 8-12 ng/ml during the first 24 weeks post-transplant and 5-8 ng/mL thereafter.
- Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept: Induction:
  Methylprednisolone (MEDROL) was administered at a dose of 500mg on the day of transplant, and tapered to 250 mg on day 1, 125 mg on day 2, 60 mg on day 3, 30 mg on day 4, and 0 mg on day 5.
  Thymoglobulin via intravenous infusion was administered at a target dose of 6 mg/kg over 3 to 4 days.
  Maintenance:
  Belatacept (NULOJIX) was given at a dose of 10 mg/kg beginning 24 hours from the time of reperfusion, and then at days 5, 14, 28, 56 and 84.
  Mycophenolate Mofetil (MMF) or equivalent was administered at a target dose of 1000 mg PO or IV BID starting on the day of transplant or day 1.
- Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept: Induction:
  Methylprednisolone (MEDROL) was administered at 500mg on day of transplant, and tapered to 250 mg on day 1, 125 mg on day 2, 60 mg on day 3, 30 mg on day 4, and 0 mg on day 5.
  Basiliximab (Simulect) was administered in two 20 mg doses, within 2 hours prior to transplantation and on day 3.
  The site investigator determined the initial tacrolimus (tac) dose started on the day of transplant or day 1. Dosing was adjusted to achieve a target trough of 8-12 ng/ml during days 1-84, and then decreased by 1/3 at day 84 and by 1/3 at week 16. If trough levels were less than or equal to 3 ng/ml at week 20 then all tac was stopped. Otherwise, the dose was reduced by 1/2 and stopped at week 24.
  Maintenance:
  Mycophenolate Mofetil (MMF) or equivalent was administered at a target dose of 1000 mg PO or IV BID starting on the day of transplant or day 1.
  Belatacept (NULOJIX) was given at 10 mg/kg beginning 24 hours from the time of reperfusion, and at days 5, 14, 28, 56 and 84
- Enrolled, Not Randomized: Subjects who signed informed consent and were thus enrolled, but were not randomized to study treatment.
Period: Overall Study
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept | Enrolled, Not Randomized
Started | 29 | 29 | 11 | 2
Completed | 26 | 28 | 11 | 0
Not Completed | 3 | 1 | 0 | 2
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Donor complication | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept | Total
Number analyzed (Participants) | 29 | 29 | 11 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 11 | 69
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (6.76) | 44.5 (10.45) | 44.6 (9.63) | 45.9 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 4 | 21
  Male | 20 | 21 | 7 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 26 | 25 | 9 | 60
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 13 | 5 | 34
  White | 9 | 11 | 4 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 11 | 69

OUTCOME MEASURES:

1. Primary Outcome: Mean Estimated Glomerular Filtration Rate (eGFR) Calculated for Each Treatment Group Using the CKD-EPI Equation at Wk 52 Post-Transplant
Description: eGFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI):
  * A score of ≥90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate very severe or end stage kidney failure.
Time Frame: Week 52
Population: Intent-to-treat population with available data at week 52
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 27 | 11
mL/min/1.73m^2 | 59.2 (19.9) | 61.5 (23.3) | 63.0 (17.4)
Statistical Analysis 1: Comparison: Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac vs Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept; Test type: Superiority; p = 0.544, Mixed Models Analysis; Mean Difference (Final Values) = 3.512, 95% CI 2-sided [-7.999 to 15.024] — The p-value, estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from weeks 4, 12, 28, 36, and 52 to compare Group 2 to Group 1
Statistical Analysis 2: Comparison: Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac vs Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept; Test type: Superiority; p = 0.531, Mixed Models Analysis; Mean Difference (Final Values) = 4.820, 95% CI 2-sided [-10.481 to 20.121] — P-value estimate of the treatment group difference, and estimated 95% confidence interval result from a repeated measures mixed model using available eGFR data from weeks 4, 12, 28, 36, and 52 to compare Group 3 to Group 1

2. Secondary Outcome: Count of Participants With Biopsy Proven Acute Rejection By Wk 52 Post-Transplant
Description: Biopsy proven acute rejection definition: histologic evidence of a Banff grade of ≥1A per local pathologist.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 1 | 10 | 4

3. Secondary Outcome: Count of Participants With eGFR < 60 mL/Min/1.73 m^2 Measured by CKD-EPI at Wk 52 Post-Transplant
Description: as for outcome 1
Time Frame: Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 21 | 15 | 6

4. Secondary Outcome: Count of Participants by CKD Stage at Wk 52
Description: The stages of Chronic Kidney Disease are defined using the participant's GFR value:
  * Stage 1 if GFR value is ≥90 ( kidney function is normal)
  * Stage 2 if 60 ≤ GFR < 90 (mildly reduced kidney function, pointing to kidney disease)
  * Stage 3A if 45 ≤ GFR < 60*
  * Stage 3B if 30 ≤ GFR < 45*
  * Stage 4 if 15 ≤ GFR < 30 (severely reduced kidney function)
  * Stage 5 if GFR < 15 (severe or end stage kidney failure).
  Stages 3A and 3B indicate moderately reduced kidney function.*
Time Frame: Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  Stage 1 | 3 | 3 | 1
  Stage 2 | 5 | 11 | 4
  Stage 3A | 11 | 9 | 6
  Stage 3B | 6 | 2 | 0
  Stage 4 | 1 | 1 | 0
  Stage 5 | 3 | 3 | 0

5. Secondary Outcome: Count of Participants With Defined CKD Stage 4 or 5 at Wk 52 Post-Transplant
Description: The stages of Chronic Kidney Disease (CKD) are defined using the participant's GFR value:
  * Stage 1 if GFR value is ≥ 90 (kidney function is normal)
  * Stage 2 if 60 ≤ GFR < 90 (mildly reduced kidney function, pointing to kidney disease)
  * Stage 3A if 45 <= GFR < 60*
  * Stage 3B if 30 <= GFR < 45*
  * Stage 4 if 15 ≤ GFR < 30 (severely reduced kidney function)
  * Stage 5 if GFR < 15 (severe or end stage kidney failure).
  Stages 3A abd 3B indicate moderately reduced kidney function.*
Time Frame: Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 4 | 4 | 0

6. Secondary Outcome: Mean Calculated eGFR Using MDRD 4 Variable Model at Wk 52 Post-Transplant
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Modification of Diet in Renal Disease equation (MDRD):
  * A score of ≥ 90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate severe or endstage kidney failure.
Time Frame: Week 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 27 | 11
mL/min/1.73m^2 | 56.1 (18.5) | 57.0 (20.7) | 58.2 (14.4)

7. Secondary Outcome: The Slope of eGFR by CKD-EPI Over Time Based on Serum Creatinine Post-Transplant
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI):
  * A score of ≥ 90 means kidney function is normal.
  * A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease.
  * Scores between 30 and 59 indicates moderately reduced kidney function.
  * Scores between 15 and 29 indicate severely reduced kidney function.
  * Scores below 15 indicate very severe or endstage kidney failure.
  An estimate of the slope, or change over time, in eGFR was produced using standard statistical linear modeling procedures. The estimate was then re-scaled so that it could be interpreted as a change in eGFR per month. Positive numbers indicate increasing kidney function.
  Larger numbers indicate greater change in kidney function.
Time Frame: Day 28 through Week 52 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: eGFR change over time (by month)
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 28 | 29 | 11
eGFR change over time (by month) | 0.3 (4.1) | 1.3 (2.6) | 0.8 (1.4)

8. Secondary Outcome: Count of Participants With Delayed Graft Function at Wk 52 Post-Transplant
Description: Delayed grafted function is defined as dialysis in the first week on one or more occasions for any indication other than the treatment of acute hyperkalemia in the setting of otherwise acceptable renal function.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 6 | 9 | 0

9. Secondary Outcome: Count of Participants With Acute Cellular Rejection Grade ≥ IA Defined by Banff 2007 Criteria By Wk 52 Post-Transplant
Description: Acute cellular rejection occurs when lesions at the site of the graft characteristically are infiltrated with large numbers of lymphocytes and macrophages that cause tissue damage. Acute cellular rejection for this endpoint is defined as a grade equal to or greater than IA by Banff 2007 criteria as determined by local pathology.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 1 | 10 | 4

10. Secondary Outcome: Count of Participants by Severity of First Acute Cellular Rejection by Wk 52 Post-Transplant
Description: Acute cellular rejection occurs when lesions at the site of the graft characteristically are infiltrated with large numbers of lymphocytes and macrophages that cause tissue damage. Acute cellular rejection for this endpoint is defined as a grade equal to or greater than IA by Banff 2007 criteria as determined by local pathology. Severity is graded as IA, IB, IIA, IIB, or III, with IA being the mildest form of cellular rejection and III being the most severe form of cellular rejection. Originally it was 2 endpoints but all participants' highest grade was also their first grade so only reporting their first grade.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  IA | 0 | 3 | 2
  IB | 1 | 1 | 2
  IIA | 0 | 4 | 0
  IIB | 0 | 0 | 0
  III | 0 | 2 | 0

11. Secondary Outcome: Count of Participants With Antibody Mediated Rejection by Wk 52 Post-Transplant
Description: Antibody mediated rejection is defined by diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury and was determined by local pathology.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 1 | 1 | 0

12. Secondary Outcome: Type of Rejection Classified by Pathologist - For Cause Kidney Biopsies
Description: Upon having a biopsy performed, persons often receive treatment for rejection based on the results of the biopsy, which may or may not have shown signs of rejection. Details of local biopsy findings are presented here for rejection. Acronyms and abbreviations are defined as follows:
  * ACR= Acute T-Cell Mediated rejection
  * AMR= Acute Antibody-mediated rejection
  * Chr. AMR=Chronic Antibody Mediated Rejection
  * Gd.=Grade
  * IFTA=Interstitial Fibrosis and Tubular Atrophy
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Number; unit: Biopsy
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Biopsy
  Borderline | 3 | 5 | 0
  Borderline, AMR-Gd. I (ATN-Like) | 1 | 0 | 0
  Borderline, AMR-Gd.I (ATN-Like), Chr.AMR, IFTA-Gd1 | 1 | 0 | 0
  Borderline, AMR-Gd. I (ATN-Like), IFTA-Gd. I | 0 | 1 | 0
  Borderline, Chr.AMR, IFTA-Gd. I | 1 | 0 | 0
  Borderline, IFTA-Gd. I | 1 | 2 | 1
  Borderline, IFTA- Gd. II | 2 | 1 | 0
  ACR-Gd. IA | 0 | 4 | 2
  ACR-Gd. IA, IFTA-Gd. I | 0 | 1 | 0
  ACR-Gd. IA, IFTA-Gd. II | 1 | 0 | 0
  ACR-Gd. IB | 1 | 0 | 0
  ACR-Gd. IB, IFTA-Gd. I | 0 | 1 | 1
  ACR-Gd. IB, IFTA-Gd. II | 0 | 0 | 1
  ACR-Gd. IB, IFTA-Gd. III | 0 | 1 | 0
  ACR-Gd. IIA | 0 | 2 | 0
  ACR-Gd. IIA, IFTA-Gd. I | 0 | 2 | 0
  ACR-Gd. III | 0 | 2 | 0
  AMR-Gd. II (Capillary/Glomerular) | 1 | 0 | 0
  IFTA-Gd. I | 4 | 5 | 1
  IFTA-Gd. II | 1 | 2 | 0

13. Secondary Outcome: Type of Treatment for Detected Graft Rejection
Description: Upon having a biopsy performed, persons often receive treatment for rejection based on the results of the biopsy, which may or may not have shown signs of rejection. Details of treatment are presented here for rejection. Acronyms and abbreviations are defined below.
  ATG=Thymoglobulin
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Number; unit: Biopsy
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Biopsy
  ATG | 0 | 1 | 0
  ATG, Pulse Steroids | 0 | 5 | 2
  ATG, Pulse Steroids, Prograf | 0 | 1 | 0
  Antibiotic | 1 | 0 | 0
  Plasmapheresis | 1 | 0 | 0
  Plasmapheresis, Oral Steroids | 1 | 0 | 0
  Pulse Steroids | 6 | 9 | 3
  Pulse Steroids, Leflunomide | 0 | 1 | 0
  Pulse Steroids, Plasmapheresis, Eculizumab | 1 | 0 | 0
  Prednisone | 0 | 2 | 0

14. Secondary Outcome: Count of Participants With De Novo Anti-Donor Histocompatibility Antigen (HLA) Antibodies at Wk 52 Post-Transplant
Description: The presence of antibodies reactive to Histocompatibility Antigen (HLA) molecules expressed on the renal allograft have been associated with both acute and chronic injury to the transplanted kidney. The development of de novo anti donor HLA antibodies may mean a person is more likely to reject the graft.
  No data available.
Time Frame: Week 52
Population: No analysis due to no available data. Data were not reported from the central laboratory and, therefore, unable to be summarized.
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Count of Participants With Either New Onset Diabetes After Transplant (NODAT) or Impaired Fasting Glucose (IFG) at Week 52 Post-Transplant -Based on Criteria Specified by the ADA and WHO
Description: New onset diabetes is the development of diabetes post-kidney transplant. It was identified by the clinical sites caring for each participant and reported directly in the clinical database. Impaired fasting glucose (IFG) is a determination made by referencing glucose measurements obtained from a standard chemistry panel. Any fasting glucose measure that is between 110 and 125 mg/dL is classified as IFG.
  Acronyms: American Diabetes Association (ADA); World Health Organization (WHO).
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  New onset diabetes during first 52 weeks | 1 | 1 | 0
  Impaired fasting glucose at week 52: number analyzed (Participants) | 14 | 15 | 8
  Impaired fasting glucose at week 52 | 2 | 0 | 0

16. Secondary Outcome: Count of Participants With Treated Diabetes Between Day 14 and Wk 52 Post-Transplant
Description: Treated diabetes is defined as receipt of any oral medication or insulin for the treatment of diabetes for >14 days.
Time Frame: Day 14 through week 52
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 28 | 11
Participants | 3 | 2 | 0

17. Secondary Outcome: Hemoglobin A1c (HbA1c) Measurements Over Time
Description: Hemoglobin A1c (HbA1c) measures the average blood glucose levels over 8-12 weeks, thus acting as a useful long-term gauge of blood glucose control:
  * A value below 6.0% reflects normal levels,
  * 6.0% to 6.4% reflects prediabetes, and
  * a value of ≥ 6.5% reflects diabetes.
Time Frame: Baseline (Pre-Transplant) and Days 28 and -84, and Weeks 28, -36, and -52 Post-Transplant
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 28 | 11
percentage
  Baseline: number analyzed (Participants) | 26 | 28 | 10
  Baseline | 5.7 (1.3) | 5.7 (1.1) | 5.9 (0.8)
  Day 28: number analyzed (Participants) | 25 | 27 | 11
  Day 28 | 5.4 (0.8) | 5.6 (1.0) | 5.4 (1.1)
  Day 84: number analyzed (Participants) | 24 | 24 | 11
  Day 84 | 5.6 (1.1) | 5.5 (1.1) | 5.4 (0.8)
  Week 28: number analyzed (Participants) | 20 | 17 | 11
  Week 28 | 6.2 (1.9) | 6.0 (1.4) | 5.6 (0.8)
  Week 36: number analyzed (Participants) | 15 | 15 | 11
  Week 36 | 6.7 (2.6) | 5.9 (1.2) | 5.5 (0.8)
  Week 52: number analyzed (Participants) | 10 | 9 | 9
  Week 52 | 7.8 (3.3) | 6.7 (1.6) | 5.8 (1.3)

18. Secondary Outcome: Standardized Blood Pressure Measurement at Wk 52 Post-Transplant
Description: A blood pressure measurement consists of two numbers: the systolic and diastolic pressures. Systolic pressure measures the pressure in blood vessels when the heart beats. Diastolic pressure measures the pressure in blood vessels between beats of the heart.
  * Systolic measures of <120 and diastolic measures of <80 are considered normal.
  * Systolic measures of 120-139 and diastolic measures of 80-89 are considered at risk (or pre-hypertension).
  * Systolic measures of ≥140 and diastolic measures of ≥90 are considered high.
Time Frame: Week 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 18 | 3
mmHg
  Systolic BP at W52 | 135.0 (18.9) | 133.7 (14.7) | 132.0 (8.7)
  Diastolic BP at W52 | 77.7 (10.9) | 79.1 (10.2) | 75.7 (13.1)

19. Secondary Outcome: Count of Participants With Use of Anti-hypertensive Medication at Wk 52 Post-Transplant
Description: Anti-hypertensive medications are a class of drugs that are used to treat hypertension. The medications seek to prevent the complications of high blood pressure, such as stroke and myocardial infarction.
Time Frame: Week 52
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 26 | 28 | 11
Participants | 18 | 23 | 8

20. Secondary Outcome: Fasting Lipid Profile at Baseline (Pre-Transplant)
Description: A fasting lipid profiles measures total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels. These measurements are used in assessing one's risk of cardiovascular disease. Target ranges for each of these measures are provided:
  * Total cholesterol: 75-169 mg/dL if age ≤20; 100-199 mg/dL if age ≥ 21; high values indicate risk of cardiovascular disease
  * LDL cholesterol: <70 mg/dL for people with documented cardiovascular disease or metabolic syndrome; <100 mg/dL for people considered high risk for cardiovascular disease; <130 mg/dL for people considered low risk for cardiovascular disease; high values indicate risk of cardiovascular disease
  * HDL cholesterol: 40mg/dL and higher; high values indicate reduced risk of cardiovascular disease
  * Non-HDL cholesterol: 30 mg/dL above the target value for LDL cholesterol; high values indicate risk of cardiovascular disease and
  * Triglycerides: <150 mg/dL; high values indicate risk of cardiovascular disease.
Time Frame: Baseline
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 22 | 26 | 7
mg/dL
  Total cholesterol | 167.1 (37.5) | 159.4 (45.0) | 167.6 (84.8)
  Non-HDL | 122.0 (35.1) | 116.1 (45.7) | 123.4 (85.3)
  LDL: number analyzed (Participants) | 21 | 25 | 6
  LDL | 91.1 (28.0) | 83.1 (38.5) | 65.2 (15.3)
  HDL | 45.1 (11.8) | 43.3 (13.0) | 44.1 (19.9)
  Triglyceride | 156.8 (103.6) | 194.4 (171.1) | 227.1 (248.1)

21. Secondary Outcome: Fasting Lipid Profile at Wk 28 Post-Transplant
Description: as for outcome 20
Time Frame: Week 28
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 15 | 15 | 10
mg/dL
  Total cholesterol | 169.6 (38.6) | 179.5 (44.4) | 167.3 (39.5)
  Non-HDL: number analyzed (Participants) | 14 | 15 | 10
  Non-HDL | 119.6 (35.9) | 133.5 (46.7) | 115.0 (38.0)
  LDL: number analyzed (Participants) | 14 | 14 | 10
  LDL | 95.6 (31.4) | 109.8 (43.0) | 82.7 (18.2)
  HDL: number analyzed (Participants) | 14 | 15 | 10
  HDL | 51.0 (14.5) | 46.0 (18.6) | 52.3 (27.5)
  Triglyceride: number analyzed (Participants) | 14 | 15 | 10
  Triglyceride | 126.4 (51.0) | 153.3 (93.0) | 166.6 (128.9)

22. Secondary Outcome: Fasting Lipid Profile at Wk 52 Post-Transplant
Description: A fasting lipid profiles measures total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels. These measurements are used in assessing one's risk of cardiovascular disease. Target ranges for each of these measures are provided:
  * Total cholesterol: 75-169 mg/dL if age ≤ 20; 100-199 mg/dL if age ≥ 21; high values indicate risk of cardiovascular disease
  * LDL cholesterol: <70 mg/dL for people with documented cardiovascular disease or metabolic syndrome; <100 mg/dL for people considered high risk for cardiovascular disease; <130 mg/dL for people considered low risk for cardiovascular disease; high values indicate risk of cardiovascular disease
  * HDL cholesterol: 40mg/dL and higher; high values indicate reduced risk of cardiovascular disease
  * Non-HDL cholesterol: 30 mg/dL above the target value for LDL cholesterol; high values indicate risk of cardiovascular disease and
  * Triglycerides: <150 mg/dL; high values indicate risk of cardiovascular disease.
Time Frame: Week 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 8 | 9 | 8
mg/dL
  Total cholesterol | 177.1 (25.6) | 163.7 (38.8) | 174.8 (54.7)
  Non-HDL | 128.6 (30.6) | 121.2 (32.0) | 130.8 (45.6)
  LDL | 102.9 (17.7) | 86.3 (50.6) | 94.6 (46.4)
  HDL | 48.5 (11.3) | 42.4 (15.6) | 44.0 (14.9)
  Triglyceride | 125.8 (93.0) | 170.0 (118.6) | 182.8 (84.2)

23. Secondary Outcome: Count of Participants With Use of Lipid Lowering Medications at Baseline and Wk 28 and Wk 52 Post-Transplant
Description: Lipid lowering medications are used in the treatment of high levels of fats (lipids), such as cholesterol in blood.
Time Frame: Baseline (Pre-Transplant), Week 28, and Week 52
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  Baseline | 13 | 7 | 3
  Week 28: number analyzed (Participants) | 27 | 29 | 11
  Week 28 | 8 | 9 | 4
  Week 52: number analyzed (Participants) | 26 | 28 | 11
  Week 52 | 9 | 9 | 5

24. Secondary Outcome: Total Daily Prescribed Pill Count
Description: This is a measure of the total number of pills a participant was prescribed on a given day
Time Frame: Day 28, Day 84, Week 28, Week 36, and Week 52
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: pills per day
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 28 | 28 | 11
pills per day
  Day 28 | 25.8 (9.9) | 18.9 (7.5) | 23.5 (8.9)
  Day 84: number analyzed (Participants) | 25 | 26 | 11
  Day 84 | 22.2 (6.3) | 17.2 (6.3) | 21.0 (7.0)
  Week 28: number analyzed (Participants) | 19 | 17 | 11
  Week 28 | 19.7 (7.2) | 15.5 (6.0) | 16.6 (8.1)
  Week 36: number analyzed (Participants) | 13 | 14 | 11
  Week 36 | 19.1 (8.0) | 15.4 (4.8) | 13.9 (5.9)
  Week 52: number analyzed (Participants) | 7 | 9 | 9
  Week 52 | 24.4 (11.8) | 15.7 (5.4) | 13.7 (5.1)

25. Secondary Outcome: Count of Participant Deaths or Graft Loss by Wk 52 Post-Transplant
Description: This measure counts deaths and graft loss occurring at any point post transplantation. Graft loss is defined as 90 days of dialysis dependency.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 2 | 0 | 0

26. Secondary Outcome: Count of Participants With Graft Rejection by Wk 52 Post-Transplant
Description: The number of participants who were treated by their local physician for any type of rejection including, but not limited to cellular rejection and antibody- mediated rejection of the transplanted kidney regardless of the presence of a biopsy.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 7 | 14 | 4

27. Secondary Outcome: Count of Participants Experiencing ≥ 1 Adverse Event (AEs) or Serious Adverse Events (SAEs) by Wk 52
Description: Adverse events were collected systematically from enrollment through Wk 52, the last study visit. Provided are numbers of participants with ≥ 1 adverse event (serious or non-serious adverse events) by treatment arm.
Time Frame: Enrollment through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  Adverse Events | 21 | 28 | 9
  Serious Adverse Events | 19 | 21 | 6

28. Secondary Outcome: Count of Participants With Infections Requiring Hospitalization or Systemic Therapy by Wk 52 Post-Transplant
Description: Infections of certain types (i.e., excluding those identified in the protocol as occurring commonly in this study population) were required to be reported as a serious adverse event if they required either inpatient hospitalization or prolongation of a current hospitalization.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 1 | 8 | 2

29. Secondary Outcome: Count of Participants With BK Polyoma Virus (BKV) and Cytomegalovirus (CMV) Viremia (Local Center Monitoring) as Adverse Events by Wk 52 Post-Transplant
Description: Viral infections following renal transplantation is significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss. Specific viruses were monitored during the study, using participant blood samples. Displayed are counts of participants who experienced BKV and CMV viremia as adverse events by treatment arm.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  BKV | 0 | 4 | 1
  CMV | 1 | 6 | 1

30. Secondary Outcome: Count of Participants With Epstein-Barr Virus (EBV) Infection as Reported on the Case Report Form as Adverse Events
Description: Viral infections following renal transplantation, including but not limited to EBV infection, is a significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants | 0 | 0 | 0

31. Secondary Outcome: Count of Participants With Fever > 39 Degrees Celsius and Blood Pressure < 90 mmHg Within 24 Hours of Onset of Transplant Procedure
Description: Temperature of >39 degrees Celsius (e.g., 102.2 degrees Fahrenheit) would be an indication of fever most often in response to an infection or illness. Systolic blood pressure <90mm Hg would be an indication of low blood pressure.
Time Frame: Within 24 Hours of transplant procedure
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept
Number analyzed (Participants) | 29 | 29 | 11
Participants
  Fever >39 Celsius | 0 | 0 | 0
  Systolic BP < 90 mmHg | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (up to Week 52)
Arm/Group | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept | Enrolled, Not Randomized
All-Cause Mortality (participants affected / at risk) | 2/29 | 0/29 | 0/11 | 0/2
Serious Adverse Events (participants affected / at risk) | 19/29 | 21/29 | 6/11 | 0/2
Other Adverse Events (participants affected / at risk) | 15/29 | 24/29 | 7/11 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac (N=29) | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept (N=29) | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept (N=11) | Enrolled, Not Randomized (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 2 (2) | 8 (10) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (5) | 1 (1) | 0 (0)
Zygomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perinephric collection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal artery dissection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Tac (N=29) | Induction:MEDROL+Thymoglobulin, Maintenance:MMF+Belatacept (N=29) | Induction:MEDROL+Simulect+Tac, Maintenance:MMF+Belatacept (N=11) | Enrolled, Not Randomized (N=2)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 5 (5) | 3 (3) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (2) | 4 (6) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (3) | 8 (9) | 0 (0) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 (3) | 8 (8) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (4) | 3 (4) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (5) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No